CLINICAL TRIAL: NCT01951859
Title: A Double Blind Placebo Controlled Pilot Study to Evaluate the Effects of a Homeopathic Anti-inflammatory Topical Cream on the Healing of Wounds That Develop Into Ulcers and Neuropathy in the Diabetic Foot.
Brief Title: Effects of a Homeopathic Anti-inflammatory Topical Cream on Ulcers and Neuropathy in the Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Principal Investigator, Oscar M. Alvarez, PhD, Director, Center for Curative and Palliative Wound Care, Calvary Hospital, Bronx, NY
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUC-DERM-0213-DFU
Record Dates: First submitted 2013-09-16; First posted 2013-09-27 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Neuropathy/Ulcer Cream (Experimental): an anti-inflammatory topical cream that contains homeopathic ingredients
  Interventions: Other: Neuropathy/Ulcer Homeopathic topical cream
- Placebo Cream (Placebo Comparator)

INTERVENTIONS:
Other: Neuropathy/Ulcer Homeopathic topical cream — This is a GRAS topical agent containing homeopathic ingredients
  Other Names: Nan's Cream
  Arms: Topical Neuropathy/Ulcer Cream

SUMMARY:
This is a study whose primary objective is to assess the effectiveness of Neuropathy/Ulcer Cream in the promotion of healing skin fissures plantar foot ulcers and as a moisturizer to prevent dry skin turning into ulcers as compared with a placebo cream containing the same vehicle as Neuropathy/Ulcer Cream without the active ingredients (Control).

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient is 18 years old or older.

  2. Patient has a current diagnosis of diabetes (Type 1 or 2).

  3. Patient's fissure or foot ulcer is on the plantar surface of the foot.

  4. Patient's fissure or ulcer is at least a partial thickness wound extending through the epidermis and at least part of the dermis. The wound may extend through the dermis and into subcutaneous tissue (granulation tissue may be present), but without exposure of muscle, tendon, bone, or joint capsule (Wagner Grade 1).

  5. Patient's wound is free of necrotic debris and clinical infection, should be comprised of healthy, vascular tissue.

  6. Patient's Ankle-Brachial Index (ABI) by Doppler is 0.7.

  7. The patient has adequate circulation to the foot to allow for healing.

This must be demonstrated by either of the following methods:

The patient has a palpable pulse on the study foot (either dorsalis pedis, posterior tibial, or peroneal artery) and has clinical signs of adequate circulation in the foot (e.g., toes are warm and pink).

If either there are no palpable pulses or clinical signs of adequate circulation are lacking, the Investigator must perform an additional assessment to assure that there is adequate circulation to the foot. Transcutaneous oxygen tension (TcPo2), photoplethysmography (PPG), Toe-Arm Index, Doppler wave form, Cardiosynchronous Limb Compression (CSC), Pulse Volume Recording (PVR) or exercise Ankle-Brachial Index (ABI). Determination of adequate circulation must be according to generally accepted criteria for the particular test employed. The additional assessments must be documented in the patient's source document and Case Report Form.

8. Patient's diabetes is under control as determined by the Investigator from daily glucometer diary entries.

9. Patient and caregiver are willing to participate in the clinical study and can comply with the follow-up regimen.

10.Patient or his/her legal representative has read and signed the Institutional Review Board (IRB) approved Informed Consent form before treatment.

Exclusion Criteria:

1. Patient has clinical evidence of gangrene on any part of the affected foot.
2. The patient's ulcer is due to a nondiabetic etiology. Ulcers of arterial, venous stasis, pressure, radiation, traumatic, rheumatoid, vasculitis, collagen vascular disease,or other nondiabetic etiologies are not to be enrolled.
3. Patient's ulcer has tunnels or sinus tracts that cannot be completely debrided.
4. Patient's diabetes is uncontrolled and could interfere with the completion of the study.
5. Patient has one or more medical condition(s), including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the Investigator would make the patient an inappropriate candidate for this wound healing study.
6. Patient has or has had a malignant disease (other than cutaneous epithelioma) not in remission for five years or more.
7. Patient is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents, or is anticipated to require such agents during the course of the study.
8. Patient has Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV).
9. Patient has participated in another study utilizing an investigational drug or device within the previous 30 days.
10. Patient's ulcer is infected or accompanied by active cellulitis, osteomyelitis as determined by the investigator
11. Patient has any condition(s) that seriously compromises the patient's ability to complete this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-01 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Decrease in area or closure of wounds/fissures due to Homeopathic Anti-inflammatory Topical Cream | 12 weeks or wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, PhD, Principal Investigator — Wound Care Cenetr Calvary Hospital, Bronx, NY; Martin Wendelken, RN, DPM, Study Director — Podiatrist, Wound care center Calvary Hospital, Bronx, NY
Locations (1):
- Calvary Hospital Wound Care Clinic, The Bronx, New York, United States